CLINICAL TRIAL: NCT03438227
Title: Intravenous Iron for Iron-deficiency Anemia in Pregnancy: a Randomized Controlled Trial
Acronym: IVIDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Method Tuuli, Professor of Obstetrics and Gynecology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1809251633
Record Dates: First submitted 2018-01-25; First posted 2018-02-19 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Iron Deficiency Anemia of Pregnancy; Iron Malabsorption
Keywords: Iron Deficiency Anemia of Pregnancy; oral iron supplementation; parenteral iron supplementation; maternal anemia
MeSH Terms: interventions — Iron-Dextran Complex; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: All participants at less than 28 weeks gestation will have an anemia evaluation and work up per standard prenatal care. Those who meet a clinical diagnosis of iron-deficiency anemia will initiate oral iron and have their Complete Blood Count rechecked between 24 and 28 weeks gestation. If their hemoglobin is less than 10 mg/dL, they will be randomized to either continue their oral iron supplementation or receive a single intravenous dextran iron transfusion. If the patient is enrolled after 28 weeks and receives a diagnosis of iron deficiency anemia, she will be randomized at that time.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research team will be blinded to the patients' treatment arm. A team of resident physicians who are unfamiliar with the study aims will provide standard obstetric care to all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous iron dextran infusion (Experimental): Women randomized to receive intravenous iron infusion will receive a single infusion of dextran 1000mg IV as an inpatient on the antepartum or Labor & Delivery Unit. They will receive continuous fetal monitoring for 30 minutes before and after the infusion as well for the duration of the infusion
  Interventions: Drug: Iron dextran
- Oral ferrous sulfate supplementation (Active Comparator): Women randomized to continue oral iron will continue to take ferrous sulfate 325mg one to three tablets daily, with the final dose at the discretion of the patient's obstetric provider.
  Interventions: Drug: Ferrous sulfate 325mg

INTERVENTIONS:
Drug: Iron dextran — Single intravenous infusion of iron dextran 1000mg.
  Other Names: Experimental
  Arms: Intravenous iron dextran infusion
Drug: Ferrous sulfate 325mg — Oral iron supplementation with ferrous sulfate 325mg one to three times daily
  Other Names: Active comparator
  Arms: Oral ferrous sulfate supplementation

SUMMARY:
Iron deficiency is the most common cause of anemia in pregnancy worldwide, and, when severe, can have serious consequences for mothers and babies. While treatment of iron-deficiency anemia with iron supplementation is recommended, treatment strategies remain controversial: the American College of Obstetrics and Gynecology recommends oral iron supplementation with parental iron reserved for the rare patient who cannot tolerate or will not take oral iron, while United Kingdom professional organizations recommend a more liberal use of parenteral iron. The reason for these disparate recommendations is that few high-quality studies comparing oral to parenteral iron have been conducted in developed countries, and the potential impact of parental iron treatment on obstetric and perinatal outcomes remains unclear. We propose the first randomized-controlled trial in the United States describing the effectiveness and safety of treating pregnant women with iron-deficiency anemia with a protocol including parenteral iron compared with a protocol based on oral iron.

DETAILED DESCRIPTION:
Iron deficiency is the most common cause of anemia in pregnancy worldwide, and, when severe, can have serious consequences for mothers and babies. In the United States, anemia affects nearly 20% of pregnancies and the majority is iron-deficiency anemia. Therefore, treatment of iron-deficiency anemia with iron supplementation is recommended.1 However, there is controversy about the treatment strategies.

The American College of Obstetrics and Gynecology recommends oral iron supplementation for iron-deficiency anemia in pregnancy, with parental iron reserved only for the "rare patient who cannot tolerate or will not take oral iron" (1) Conversely, guidelines from the United Kingdom. are more liberal on the use of parental iron for the treatment of iron-deficiency anemia in pregnancy (2). Both treatment guidelines are based on limited data regarding the risks and benefits of parental iron for treatment of iron-deficiency anemia in pregnancy. The majority of randomized trials were conducted in developing country settings. In fact, few high-quality studies have been conducted in developed countries, and none has been conducted in the United States Moreover, there is limited data from prior studies on the impact of parental iron treatment on perinatal outcomes. The most recent Cochrane review including mostly from trials conducted in low-income countries found that, although parenteral iron improved hemoglobin levels and iron stores than the oral route, no clinical outcomes were assessed and there were insufficient data on adverse effects (3). The authors concluded that "large, good quality trials, assessing clinical outcomes including adverse effects … are required" (3).

This randomized controlled trial aims to assess the effectiveness and safety of treating pregnant women with iron-deficiency anemia with a protocol including parenteral iron compared with a protocol based on oral iron. We hypothesize that treating iron-deficiency anemia with parental iron is associated with improved maternal and neonatal outcomes compared with a protocol based on oral iron. To increase generalizability of the findings, we will use broad inclusion criteria and analyze data using the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Iron-deficiency anemia (serum ferritin <30 micrograms, normal hemoglobin electrophoresis, and hemoglobin <10 mg/dL), planned delivery at Barnes-Jewish Hospital

Exclusion Criteria:

* Non-iron-deficiency anemia, multiple gestation, prenatally diagnosed major fetal anomalies, known aneuploidy, planned delivery at other hospital, inability to obtain consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patients must be pregnant in order to participate
Enrollment: 38 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Method Tuuli, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Center for Outpatient Health, Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin No. 95: anemia in pregnancy. Obstet Gynecol. 2008 Jul;112(1):201-7. doi: 10.1097/AOG.0b013e3181809c0d. Erratum In: Obstet Gynecol. 2020 Jan;135(1):222. doi: 10.1097/AOG.0000000000003624. PMID 18591330
- [Background] Pavord S, Myers B, Robinson S, Allard S, Strong J, Oppenheimer C; British Committee for Standards in Haematology. UK guidelines on the management of iron deficiency in pregnancy. Br J Haematol. 2012 Mar;156(5):588-600. doi: 10.1111/j.1365-2141.2011.09012.x. PMID 22512001
- [Background] Reveiz L, Gyte GM, Cuervo LG, Casasbuenas A. Treatments for iron-deficiency anaemia in pregnancy. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD003094. doi: 10.1002/14651858.CD003094.pub3. PMID 21975735
- [Derived] Lewkowitz AK, Stout MJ, Cooke E, Deoni SC, D'Sa V, Rouse DJ, Carter EB, Tuuli MG. Intravenous versus Oral Iron for Iron-Deficiency Anemia in Pregnancy (IVIDA): A Randomized Controlled Trial. Am J Perinatol. 2022 Jun;39(8):808-815. doi: 10.1055/s-0041-1740003. Epub 2021 Nov 28. PMID 34839481

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Started | 20 | 18
Completed | 10 | 13
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [25 to 28] | 28 [21 to 32] | 28 [22 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23
Chronic hypertension [Count of Participants; unit: Participants] | 2 | 3 | 5
Prepregnancy diabetes [Count of Participants; unit: Participants] | 1 | 1 | 2
Nulliparous [Count of Participants; unit: Participants] — Patients having first birth
  Participants | 1 | 3 | 4
Prior preterm birth (<37 weeks' gestation) [Count of Participants; unit: Participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maternal Anemia at Delivery
Description: Number of participants with maternal hemoglobin <11g/dl at delivery
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
Participants | 4 | 11
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.039, Chi-squared

2. Secondary Outcome: Maternal Hemoglobin at Delivery
Description: Maternal hemoglobin on admission to inpatient obstetrics unit for delivery
Time Frame: On admission to inpatient obstetrics unit for delivery
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
g/dL | 11.0 (0.7) | 9.9 (1.1)
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.019, t-test, 2 sided

3. Secondary Outcome: Number of Participants With Medication Adverse Events
Description: Participants reporting symptoms when contacted by via telephone 2 - 3 days after their infusion of intravenous iron or initiation of oral iron
Time Frame: 2 - 3 days after single intravenous iron infusion or initiation of oral iron
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
Participants
  Severe | 0 | 0
  Mild/moderate | 3 | 3
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.029, Fisher Exact

4. Secondary Outcome: Maternal Hemoglobin Below 10g/dl at Delivery
Description: Number of participants with hemoglobin below 10g/dl at delivery
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
Participants | 1 | 7
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.029, Fisher Exact

5. Secondary Outcome: Maternal Ferritin at Delivery
Description: Maternal serum ferritin level in μg/L at delivery
Time Frame: At delivery
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
μg/L | 129.8 (117.2) | 26.6 (14.6)
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.19, t-test, 2 sided

6. Secondary Outcome: Number of Participants Who Received Blood Transfusion
Description: Participant receiving transfusion of packed red blood cells during admission for delivery of infant obtained via medical chart review.
Time Frame: During inpatient admission for delivery of neonate
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
Participants | 0 | 2
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.194, Fisher Exact

7. Secondary Outcome: Mode of Delivery
Description: Whether infant was delivered vaginally or via cesarean section
Time Frame: Once, at infant delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
Participants
  Vaginal delivery | 4 | 8
  Cesarean delivery | 6 | 5
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.414, Chi-squared

8. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age in weeks at delivery
Time Frame: Once, at infant delivery
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
weeks | 38.1 (1.0) | 36.9 (2.3)
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.15, t-test, 2 sided

9. Secondary Outcome: Birth Weight
Description: Neonatal weight at delivery
Time Frame: Obtained once, at infant delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
grams | 3174.0 (657.2) | 3029.2 (550.5)
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.571, t-test, 2 sided

10. Secondary Outcome: Umbilical Cord Arterial pH
Description: Umbilical cord arterial pH obtained at delivery
Time Frame: Drawn once from umbilical cord segment at delivery
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 9 | 13
Unitless | 7.24 (0.09) | 7.29 (0.05)
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.12, t-test, 2 sided

11. Secondary Outcome: APGAR Scores at 1 Minutes of Life
Description: The APGAR score, named after the Virginia Apgar, pediatrician who came up with it, measures the physical condition of a newborn infant on a scale ranging from a minimum of 0 (worsts) to a maximum of 10 (best).
Time Frame: Obtained at 1 minute of life
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
score on a scale | 8 [8 to 8] | 8 [8 to 8]
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.049, Log Rank

12. Secondary Outcome: Neonatal Hemoglobin
Description: Neonatal hemoglobin in g/dl at delivery
Time Frame: Drawn once from umbilical cord segment at birth
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
g/dL | 13.4 (3.4) | 13.5 (2.1)
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.933, t-test, 2 sided

13. Secondary Outcome: Composite Neonatal Morbidity (Defined by the Occurrence of One or More of 10 Neonatal Morbidities.
Description: Neonatal morbidity composite, defined by the occurrence of one or more of the following neonatal morbidities: neonatal seizures (diagnosed by clinician), intraventricular hemorrhage (diagnosed by clinician on brain MRI or Ultrasound), hypoxic-ischemic encephalopathy (diagnosed by clinician), neonatal hypothermic therapy (brain cooling as documented on inpatient record, sepsis (diagnosed by blood culture), respiratory distress syndrome (diagnosed by clinician), hyperbilirubinemia requiring photo therapy (diagnosed by clinician), birth injury (diagnosed by clinician), or meconium aspiration syndrome (diagnosed by clinician), neonatal intensive care unit admission (documented in the inpatient record).
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
Participants | 2 | 4
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.66, Fisher Exact

14. Secondary Outcome: Neonatal Ferritin
Description: Neonatal ferritin in ug/L at delivery
Time Frame: Drawn once from umbilical cord segment at birth
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
Number analyzed (Participants) | 10 | 13
ug/L | 169.4 (98.2) | 147.1 (69.2)
Statistical Analysis 1: Comparison: Intravenous Iron Dextran Infusion vs Oral Ferrous Sulfate Supplementation; Test type: Superiority; p = 0.633, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 - 3 days after the single intravenous iron infusion or initiation of oral iron
Arm/Group | Intravenous Iron Dextran Infusion | Oral Ferrous Sulfate Supplementation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 3/10 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Iron Dextran Infusion (N=10) | Oral Ferrous Sulfate Supplementation (N=13)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03438227/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03438227/ICF_001.pdf